CLINICAL TRIAL: NCT04452838
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, CROSSOVER STUDY TO ASSESS THE BIOEQUIVALENCE UNDER FED AND FASTED CONDITIONS OF FESOTERODINE BEADS-IN-CAPSULE SR7 AND SR4 FORMULATIONS, THE EFFECT OF FOOD ON THE PHARMACOKINETICS OF THE BEADS-IN-CAPSULE SR7 FORMULATION AND TO ESTIMATE THE BIOAVAILABILITY OF SR7 BEADS SPRINKLED ON APPLE SAUCE RELATIVE TO THE BEADS-IN-CAPSULE SR7 FORMULATION ADMINISTERED INTACT
Brief Title: Study To Assess The Bioequivalence Under Fed And Fasted Conditions Of The Fesoterodine Beads-In-Capsule SR4 And SR7 Formulations And To Estimate The Bioavailability of SR7 Beads Sprinkled On Apple Sauce Relative To The Beads-In-Capsule SR7 Formulation Administer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0221115; 2019-001909-24 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Phase I, Fesoterodine beads- in-capsule, Bioequivalence, Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 randomized, open-label, single-dose crossover study in healthy participants. A two stage approach outlined below will be followed:
  Part A (Cohort 1): This part of the study is a 2 sequence, 4 period, crossover design.
  Part B (Cohort 2): This part of the study is a 4 sequence, 4 period, crossover design. Participants will be randomized to 1 of 4 possible treatment sequences. If bioequivalence (BE) criteria for the comparison of the BIC SR7 formulation with the BIC SR4 formulation administered in the fasted state are met in Part A, the formulations will be considered bioequivalent in the fasted state and only the first two periods of Part B will be conducted. Part B (all periods) may not be conducted if the AUCinf or Cmax Percent Geometric Mean Ratio GMR is less than 90% and greater than 111% and/or if variability suggest a highly variable drug (e.g., greater than 30%) because BE demonstration may not be possible with a reasonably sized 4 sequence 4 period study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 Sequence 1 (Part A) (Other): Treatment Sequence A,B,C and D
  Interventions: Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B); Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B); Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B); Drug: Fesoterodine BIC SR7 on apple sauce (Treatment D in Part A)
- Cohort 1 Sequence 2 (Part A) (Other): Treatment Sequence B, A,C and D
  Interventions: Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B); Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B); Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B); Drug: Fesoterodine BIC SR7 on apple sauce (Treatment D in Part A)
- Cohort 2 Sequence 1 (Part B) (Other): Treatment Sequence E, F, G, and H
  Interventions: Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B); Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B); Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B); Drug: Fesoterodine BIC SR4 fed (Treatment E in Part B)
- Cohort 2 Sequence 2 (Part B) (Other): Treatment Sequence E, F, H and G
  Interventions: Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B); Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B); Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B); Drug: Fesoterodine BIC SR4 fed (Treatment E in Part B)
- Cohort 2 Sequence 3 (Part B) (Other): Treatment Sequence F, E, G, and H
  Interventions: Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B); Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B); Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B); Drug: Fesoterodine BIC SR4 fed (Treatment E in Part B)
- Cohort 2 Sequence 4 (Part B) (Other): Treatment sequence F, E, H, and G
  Interventions: Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B); Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B); Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B); Drug: Fesoterodine BIC SR4 fed (Treatment E in Part B)

INTERVENTIONS:
Drug: Fesoterodine BIC SR4 fasted (Treatment A in Part A, Treatment G in Part B) — 4 mg administered under fasted condition.
Drug: Fesoterodine BIC SR7 fasted (Treatment B in Part A, Treatment H in Part B) — 4 mg administered under fasted conditions.
Drug: Fesoterodine BIC SR7 fed (Treatment C in Part A, Treatment F in Part B) — 4 mg administered under fed conditions.
Drug: Fesoterodine BIC SR7 on apple sauce (Treatment D in Part A) — 4 mg sprinkled on apple sauce administered under fasting conditions
  Arms: Cohort 1 Sequence 1 (Part A); Cohort 1 Sequence 2 (Part A)
Drug: Fesoterodine BIC SR4 fed (Treatment E in Part B) — 4 mg administered under fed conditions
  Arms: Cohort 2 Sequence 1 (Part B); Cohort 2 Sequence 2 (Part B); Cohort 2 Sequence 3 (Part B); Cohort 2 Sequence 4 (Part B)

SUMMARY:
Open Label, Single-Dose, Crossover Study To Assess The Bioequivalence Under Fed And Fasted Conditions Of The Fesoterodine Beads-In-Capsule (BIC) SR4 And SR7 Formulations And To Estimate The Bioavailability of SR7 Beads Sprinkled On Apple Sauce Relative To The Beads-In-Capsule SR7 Formulation Administered Intact.

DETAILED DESCRIPTION:
After oral administration, fesoterodine is not detected in plasma as it is rapidly and extensively hydrolyzed by non-specific esterases to its primary active metabolite 5-hydroxymethyl tolterodine (5-HMT) . Therefore characterization of the rate and extent of absorption of the test and reference fesoterodine formulations will be based on pharmacokinetic parameters of 5-HMT derived from the 5-HMT concentration-time profiles.

ELIGIBILITY:
Inclusion Criteria

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures. Weight:
4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
3. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb). A positive serology for hepatitis B surface antibody (HBsAb) as a result of Hepatitis B vaccination is allowed.
4. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
5. History of allergy or hypersensitivity to fesoterodine fumarate or tolterodine tartrate, soya, or any of the excipients in the investigational drug product.
6. History of uncontrolled narrow angle glaucoma, myasthenia gravis, gastric retention, severe ulcerative colitis and toxic megacolon.
7. Evidence or history of clinically significant urologic disease: urinary retention, obstructive disturbance of bladder emptying, micturition disturbance, nocturia or pollakiuria (eg, benign prostate hyperplasia, urethral stricture, recurrent urinary tract infections).
8. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
9. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
10. A positive urine drug test, as confirmed by a single repeat.
11. Screening supine blood pressure (BP) greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
12. Screening 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is greater than 450 msec, this interval should be rate-corrected using the Fridericia method and the resulting corrected QT (QTcF) should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
13. Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:
14. Screening estimated glomerular filtration rate (eGFR) is less than or equal to 90 mL /min/1.73 m2 for Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).
15. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
16. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
17. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
18. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
AUCinf of 5-HMT | 0 (pre dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Area under the plasma concentration-time curve from time zero extrapolated to infinity.
AUClast of 5-HMT | 0 (pre dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Area under the plasma concentration-time curve from 0 to the time of the last quantifiable concentration.
Cmax of 5-HMT | 0 (pre dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Maximum Observed Plasma Concentration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A0221115